Study title: Effects of a brief parent-based sleep intervention for children with attention deficit hyperactivity disorder

Research Protocol V1.2

Date: 29th September 2016

Dated: 29<sup>th</sup> Sept, 2016 Version number: 1.2 – Clincial Trial Registration

**Background and Significance** 

Sleep disturbances as a common complaint in children with ADHD and the associated

consequences

Attention deficit hyperactivity disorder (ADHD) is the most common psychiatric disorder with

childhood onset, affecting approximately 5% of children and adolescents worldwide, and 3.9% in

Hong Kong.<sup>3</sup> It is characterized by impairment caused by inattention, impulsivity, and/or

hyperactivity. At least one comorbid psychiatric disorder is present in 87% of children with ADHD.<sup>4</sup>

Among the array of comorbidities, sleep problems and the associated impairments have long been

recognized as one of the most common issues. Sleep problems have been reported in 25-73% of

children with ADHD.<sup>5-6</sup> Local data also indicate that non-medicated ADHD children experienced

significantly more sleep difficulties than normally developing children.<sup>7</sup>

The impacts of sleep problems on ADHD children can be far-reaching. Presence of sleep problems

ranging from mild to severe predicts lower psychosocial functioning even after controlling for other

potential confounders, including comorbidities, demographic characteristics, and severity of ADHD

symptoms. 8 Moderate-to-severe sleep problems are strongly associated with the severity of ADHD

symptoms and impaired physical wellbeing of the child; parents with an ADHD child with comorbid

sleep problems are 2.7 times more likely to be clinically depressed, stressed, or anxious.<sup>6</sup>

Evidence-based treatments for sleep problems in ADHD

Within the complex and multidirectional relationship between sleep and ADHD, poor sleep hygiene

has been found to be a significant contributor. A previous study has shown that sleep problems in

ADHD are generally behavioural in nature, primarily occurring at or around sleep onset. Behavioural

interventions have been found to be effective in managing sleep problems in children in the general

population, 10 as well as in children with special needs (e.g. those with neurodevelopmental

disorders). 11-13 Hence, behavioural interventions have been suggested as the first-line treatment for

ADHD children experiencing sleep problems. 14 In fact, standard behavioural techniques, such as

graduated extinction and bedtime fading, have shown to be highly effective in managing sleep

problems in children with ADHD.<sup>10</sup>

**Significance** 

Dated: 29th Sept, 2016

Version number: 1.2 – Clincial Trial Registration

We expect that this parent-based behavioural sleep intervention will improve the sleep quality of children with ADHD, which in turn may lower inattention/hyperactivity impairment, reduce parental stress and improve the child's daily functioning.

Objectives and Hypothesis of the study

To assess the effect of a brief parent-based sleep behavioural intervention on the sleep quality as well as other aspects of functioning and mental health of children with ADHD and their parents.

Compared to children with ADHD and insomnia receiving treatment as usual, the group of children with ADHD and insomnia receiving the parent-based intervention will have better sleep and

functioning as well as parental mental health at post-intervention and follow-up at 3 months.

Study Design/Methodology

**Study Sites** 

Alice Ho Miu Ling Nethersole Hospital, TaiPo, N.T., Hong Kong

Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong

**Study Population** 

Parents of children who meet all the following inclusion criteria and none of the exclusion criteria will be our target participants.

Inclusion criteria:

ADHD with sleep problem(s)

Aged 6-12 years old;

With a clinical diagnosis of ADHD (any subtype), as confirmed by the Diagnostic
Interview Schedule for Children-version-IV (DISC-IV);

interview selledule for eliminen-version-rv (Disc-rv),

- With parent-reported insomnia (difficulty initiating sleep and/or maintaining sleep).

Exclusion criteria:

 Children with a serious medical condition (e.g. severe cerebral palsy) or intellectual disability (IQ<70);</li>

2. Children with a neurological and/or medical condition that may lead to disordered sleep;

3. Suspected clinical sleep disorders (e.g. obstructive sleep apnea, OSA) that may potentially contribute to a disruption in sleep continuity and quality, as assessed by the Children's Sleep

Habits Questionnaire (CSHQ). If the child is suspected of a clinical sleep disorder, he/she will be

Dated: 29th Sept, 2016

Version number: 1.2 – Clincial Trial Registration

referred to appropriate services;

4. Children who are already receiving specialized help for their sleep from a psychologist or at a

specialized sleep clinic.

A total of 60 families will be invited to participate in this programme and will be randomized into

intervention group and waitlist-control group (30 families each).

**Subject Recruitment Plans and Consent Process** 

Patients at the child psychiatric clinic of Alice Ho Miu Ling Nethersole Hospital who potentially meet

the inclusion criteria will be invited to take part in the study by the attending psychiatrists. Recuitment

will be also conducted in the community (e.g. via posters, mass emails).

Potential interested parents will be contacted via phone and a brief assessment will be conducted to

ascertain the presence and severity of sleep problems. For those who report that their child has

insomnia, they will be asked several questions to establish whether the problem meets the

International Classification of Sleep Disorders criteria.

Potential participants will then be invited to attend a face-to-face interview. First, consent will be

obtained from the carer/parent of the targeted child with a Cantonese consent form provided with

sufficient time for reading and enquiry. Potential participants will then be screened using CSHQ for

presence of sleep problems (exclusion criteria) and DISC-IV to further confirm the ADHD diagnosis.

Suitable participants with insomnia will then be randomized into the two groups of intervention and

wait-list control. The intervention will involve two fortnightly individual consultation sessions. The

first session will focus on (1) a thorough assessment of the nature of the child's sleep problem,

followed by (2) the provision of sleep-related psycho-education about normal sleep based on the

child's developmental level, sleep hygiene, specific strategies known to be effective in tackling

problematic sleep-related behaviours in children, and (3) collaborative goal setting and development

of management plan tailored to the child's sleep problem for the next two weeks. Parents will also be

asked to complete a sleep diary to monitor their child's sleep patterns in the following two weeks. The

second session will involve a review of the sleep diary and a reinforcement of learned strategies, and

focus on problem-solving to tackle any issues that have emerged from implementing the behavioural

strategies at home. Families will be provided with information sheets and leaflets designed for this

programme, which will include information about sleep hygiene, common sleep problems, and

strategies for managing specific sleep problems in children with ADHD. A follow-up phone call will

Dated: 29th Sept, 2016

Version number: 1.2 – Clincial Trial Registration

be made two weeks later to provide parents with an opportunity to ask any further questions and to consolidate learned strategies and further troubleshoot.

Measurements

Child-related Measures

**Sleep Problems & Daytime Functioning** 

<u>Children's Sleep Habits Questionnaire (CSHQ) – parent report.</u> A validated 50-item parentreport measure of difficulties initiating and maintaining sleep over past week in children of age 4-12

(Cronbach's alpha=0.79). Items are rated on a three-point scale from "rarely" to "usually", and scores

range from 33 to 99. The validated Chinese version will be used. 16

<u>Pediatric Daytime Sleepiness Scale (PDSS) – parent report</u>. A validated 8-item self-report

scale to measure daytime sleepiness in children and adolescents (Cronbach's Alpha=0.80). <sup>17</sup> The

Chinese version has been validated.<sup>18</sup>

Actigraphy. Assessed with Actiwatch 2 (Philips Respironics, Murrysville, PA), a small motion

sensor attached to the non-dominant wrist to measure body movements. Indicators such as total sleep

time, sleep onset latency, wake after sleep onset, and sleep efficiency (ratio of time asleep to time spent

in bed) will be measured. Movement patterns can then be analysed in terms of sleep and wake times

according to established scoring rules.<sup>19</sup>

<u>Sleep diaries – parent report</u>. Daily primary caregiver report of child sleep during the two 7-

days sessions of actigraph measurement.

**ADHD Diagnosis & Symptoms** 

Diagnostic Interview Schedule for Children – Version-IV (DISC-IV) – parent report. To

confirm the diagnosis of attention deficit/hyperactivity disorder (ADHD) based on DSM-IV.<sup>20</sup> DISC-

IV was validated locally.<sup>21</sup> Functional impairment scores to achieve a full DSM-IV diagnosis were

included, according to published scoring algorithms for the DISC-IV, equivalent to one severe or at

least two intermediate impairments in six domains of daily functioning.<sup>22</sup>

Strengths and Weaknesses of ADHD Symptoms (SWAN) – parent report. The Chinese version

of SWAN rating scale is an 18-item questionnaire for assessment of ADHD symptoms, validated locally

for Chinese children in Hong Kong.<sup>23</sup> Parents are asked to compare the child's inattention and

hyperactivity behaviours with children of the same age using a 7-point scale. Scores range from -3 (far

better than peers) to +3 (far worse than peers), with 0 denoting average behaviour. The total scale score

had excellent internal consistency (Cronbach's Alpha=0.90), test-retest reliability, and good

discriminant validity in differentiating ADHD clinic sample from community sample. <sup>23</sup>

Dated: 29th Sept, 2016

Version number: 1.2 – Clincial Trial Registration

## Behaviour, Other Clinical Symptoms & Functioning

<u>Child Behavior Checklist (CBCL) – parent report</u>. A validated 118-item measure assessing mental health problems in children and includes both externalizing and internalizing problems.<sup>24</sup> The validated Chinese version will be used.<sup>25</sup>

Pediatric Quality of Life Inventory 4.0 – parent proxy report (PedsQL) – parent report. A validated 23-item measure of quality of life for children aged 2-18 (Cronbach's alpha=0.86). A psychosocial health summary score is generated from 15 items, with scores ranging from 0 to 100 (higher scores indicating better quality of life). Items are rated on a 5-point scale from "never" to "almost always" as based on behaviour of child in the past month. A validated Chinese version by the research trust will be used (NB: the English version is attached, currently acquiring the Chinese version).

Strengths and Difficulties Questionnaire – parent report. The Strengths and Difficulties Questionnaire (SDQ) is a screening questionnaire designed by Goodman<sup>27</sup> to identify psychological maladjustment in children and adolescents. There are five domains: conduct problems, inattention-hyperactivity, emotional problems, peer problems and pro-social behaviour. Each domain contains five questions on a 3-point Likert scale. The difficulties score is the sum of all items except those on prosocial behaviour. An impact supplement scale looks at how the psychological problems of the children impact his/her surroundings. A Chinese version of SDQ is available and has proved reliable and valid.

## **Cognitive Performance**

Continuous Performance Test (CPT). <sup>29</sup>A computerised attention test designed by the Psychology Experiment Building Language, adopting the Conners Continuous Performance task (CCPT). A constant series of letter stimuli appear on the screen, participant must respond to all stimuli except for the letter X. The task takes approximately 14 minutes to complete. This task is used for measuring visual sustained attention, response inhibition, and reaction time.

<u>Digit Span</u>. <sup>30</sup> A computerised digit span task developed by the Psychology Experiment Building Language. A string of number is presented to participants both visually and auditory. Participants are then asked to key in the number string presented to them earlier. This task takes approximately 3 minutes to complete. This task is used for measuring auditory attention span.

N-back. A computerised visual working memory task, adapted from the dual n-back task designed by the Psychology Experiment Building Language. <sup>31</sup> The n-back task consists of three different load levels (1-back, 2-back, and 3-back). Continuous audio and visual information are presented to participants. Participants are asked to response to the stimulus if the target is identical to the one immediately preceding one (1-back), identical to the one presented two trails back (2-back), and identical to the one presented three trails back (3-back). It consists of 59 test trails and task takes

Dated: 29th Sept, 2016

approximately 8 minutes to complete. This task is used for measuring auditory and visual working memory.

<u>Letter-digit task</u>. <sup>32</sup> A computerized version of letter digit substitution task developed by the Psychology Experiment Building Language. Nine letters and nine digits are paired at the top of the screen and the child is requested to press the digits on the keyboard corresponding to a test set of the nine symbols presented in a mixed order. It consists of 30 trails and it takes approximately 3 minutes to complete. This task is used for measuring cognitive processing.

Bergs Card Sorting Test (BCST). <sup>33</sup> A computerised version of card sorting test adapted from Wisconsin Card Sorting Test, designed by the Psychology Experiment Building Language. BCST contains 64 screen images (cards). A number of cards are presented to the participants. Participants are asked to sort the cards depending on the particular rule. They do not know how to match, however feedback are given whether a particular match is right or wrong. This task takes approximately 3 minutes to complete. This task is used for measuring cognitive flexibility.

Tower of London (TOL). <sup>34</sup> A computerised version of the TOL task developed by the Psychology Experiment Building Language, based on Shallice (1982)<sup>35</sup> TOL paradigm. Participants are asked to move coloured discs one by one from an initial state to match a goal state, within limited moves. There are a total of 12 trails for this task. This task is used for measuring planning skills.

#### Parent-related Measures

## Sleep

<u>Pittsburgh Sleep Quality Index (PSQI)</u>. A validated 19-item measure used to assess sleep habits, quality, and quantity, producing a total score and seven sub-scores in sleep quality, sleep onset latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction (Cronbach's Alpha=0.83). <sup>36</sup> The validated Chinese version will be used. <sup>37</sup>

Insomnia Severity Index (ISI). A validated 7-item measure for detecting changes in perceived sleep difficulties, with high convergence between patient and clinician ratings (Cronbach's Alpha=0.74). <sup>38</sup> Items are rated on a 5-point scale from "not at all" to "extremely". Total score ranges from 0-28 and higher scores indicate greater insomnia severity. The Chinese version has been validated. <sup>39</sup>

<u>Sleep Hygiene Index (SHI)</u>. A validated 13-item measure designed to assess sleep hygiene (Cronbach's alpha=0.66). <sup>40</sup> Items are rated on a 5-point scale from "never" to "always". Total scores range from 0 to 52, with high scores indicating poorer sleep hygiene.

<u>Epworth Sleepiness Questionnaire (ESS)</u>. A validated 8-item measure to assess daytime sleepiness in terms of the likelihood of falling asleep while engaged in eight different activities

Dated: 29th Sept, 2016

(Cronbach's Alpha=0.74). 41 Items range from 0-3 and the total score ranges from 0-24. Higher scores indicate greater sleep propensity in daily life. The Chinese version has been validated. 42

Actigraphy. As above.

**Mental Health** 

Parental Stress Index – Short Form (PSI-SF). A validated 36-item measure on parental distress, parent-child dysfunctional interaction, and difficult child (Cronbach's Alpha=0.81). 43 The

validated Chinese version will be used. 44

<u>Depression Anxiety Stress Scales – 21 item (DASS-21)</u>. A validated 21-item measure on

adult mental health, looking at depression, anxiety, and stress (Cronbach's Alpha=0.95). 45 Items are

rated on a four-point scale from "not at all" to "most of the time", with higher scores representing

more mental health difficulties. A validated Chinese version will be used. 46

Multidimensional Fatigue Inventory (MFI). A validated 20-item measure devised to measure

fatigue; dimensions include general fatigue, physical fatigue, mental fatigue, reduced motivation, and

reduced activity (Cronbach's Alpha=0.84). 47 The Chinese version has been validated. 48

Other Information

Demographics & health history. Each family will complete a brief questionnaire so as to

provide sample characteristics of the child (demography, family characteristics, medical history).

Prescribed medication(s) of the child at the time of study will be documented and recorded.

Evaluation survey. Each family will be invited to complete a brief evaluation survey to

provide feedback on the usefulness and arrangement of the intervention.

Measures on sleep, ADHD symptoms, other clinical symptoms and functioning, and cognitive

performance of the child, as well as parental sleep and mental health will be administered at the

following time-points for the intervention and waitlist-control group: before the intervention

programme (baseline); after the intervention (one-week after the follow-up call to assess the short-

term effects of the intervention). The above measurements will be additionally conducted for the

intervention group at 3 months after the intervention to assess any long-term effects of the treatment.

**Statistical Analysis Plan** 

Sample Size Determination and Power

The primary outcome is the child's sleep based on parental report (e.g. CSHQ, sleep problems rated

by parents), as a measure of intervention efficacy. Secondary outcomes include other sleep measures

(e.g. actigraphic parameters, daytime sleepiness), daytime functioning, quality of life and other

Dated: 29th Sept, 2016

Version number: 1.2 – Clincial Trial Registration

clinical symptoms and behevaior of the child, as well as parental sleep and mental health. A previous

representative study found an effect size of -0.8 for CSHQ at 3 months follow-up, which would

require 26 families in each arm to have 80% power at the two-sided 5% level of significance to detect

this effect. <sup>49</sup> To allow for 15% loss to follow-up, we require 30 families in each group.

**Analysis Plan** 

Preliminary descriptive analysis will be conducted to compare the two groups (intervention, wait-list

control) for any baseline differences in sleep and functioning characteristics. Subsequent analysis will

be conducted on an intention to treat basis. For child- and parent-related measures, changes between

baseline and post-intervention as well as between baseline and follow-up at 3 months will be

computed. Mean differences in change at 95% confidence interval in outcomes between intervention

and control arms will be estimated with regression models, adjusting for covariates as well as baseline

scores for each specific measure if there are any group differences. <sup>50</sup> Potential covariates to be

considered include the child's age, sex, medication use (yes or no), and family socioeconomic status

(measured by monthly family income). As for computing effect sizes, changes in each outcome will

be standardized to a mean of 0 and standard deviation of 1, before repeating the regression analyses.

Effect sizes are interpreted as small, moderate and large for standard deviations of ~0.20, 0.50,

and .80 respectively. 51

**Declaration of Helsinki** 

The study will follow the ethical principles under the Declaration of Helsinki. The right of all

individuals to self-determination and the right to make informed decisions regarding participation in

research, both initially and during the course of the research are respected. Participants' welfare would

take precedence over the interests of science and society, and ethical consideration would take

precedence over laws and regulations.

**Privacy and confidentiality** 

Participants' names will be kept on a password-protected database and will be linked only with a study

identification number for this research. There are no patient identifiers. Data will be stored in a locked

office of the investigators and maintained for a minimum of three years after the completion of the

study.

Risk/Benefit to participants

This study does not present any risks to the participants. Selected participants will all receive a

behavioural sleep intervention and related education materials.

Version number: 1.2 – Clincial Trial Registration

#### References

- Clinical practice guidelines: diagnostic and evaluation of the child with attention deficit/hyperactivity disorder. American Academy of Pediatrics Committee on Quality Improvement. Pediatrics 2000; 105, 1158-1170.
- 2. Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry 2007; 164:942-8.
- 3. Leung PWL, Hung SF, Ho TP, Lee CC, Liu WS, Tang. CP, Kwong SL. Prevalence of DSM-IV disorders in Chinese adolescents and the effects of an impairment criterion. A pilot community study in Hong Kong. Eur Child Adolesc Psychiatry 2008; 17, 452–461.
- 4. Hodgkins P, Setyawan J, Mitra D, Davis K, Quintero J, Fridman M, Shaw M, Harpin V. Management of ADHD in children across Europe: patient demographics, physician characteristics and treatment patterns. Eur J Pediatr 2013; 172:895–906.
- 5. Hvolby A. Associations of sleep disturbance with ADHD: implications for treatment. ADHD Attention Deficit and Hyperactivity Disorders 2015; 7(1):1-8.
- 6. Sung V, Hiscock H, Sciberras E, Efron D. Sleep problems in children with attention-deficit/hyperactivity disorder: prevalence and the effect on the child and family. Archives of Pediatrics & Adolescent Medicine 2008; 162(4):336-42.
- Lee MMC. Sleep-problems in Hong Kong Chinese children with Attention deficit/Hyperactivity Disorder – a cross-sectional study. 2012. (Unpublished dissertation). The Hong Kong College of Psychiatrists.
- 8. Becker, S. P., Langberg, J. M., & Evans, S. W. (2015). Sleep problems predict comorbid externalizing behaviors and depression in young adolescents with attention-deficit/hyperactivity disorder. European child & adolescent psychiatry, 24(8), 897-907.
- 9. Sung V, Hiscock H, Sciberras E, Efron D. Sleep problems in children with attention-deficit/hyperactivity disorder Prevalence and the effect on the child and family. Arch Pediatr Adolesc Med 2008, 162:336-42.
- Mindell JA, Owens JA. A Clinical Guide to Pediatric Sleep: Diagnosis and Management of Sleep Problems (3<sup>rd</sup> ed.). 2015. Philadelphia: Wolters Kluwer.
- Kodak T, Piazza CC: Assessment and behavioural treatment of feeding and sleeping disorders in children Autism Spectrum Disorders. Child Adolesc Psychiatr Clin N Am 2008, 17:887-905
- 12. Montgomery P, Stores G, Wiggs L: The relative efficacy of two brief treatments for sleep problems in young learning disabled (mentally retarded) children: a randomised controlled trial. Arch Dis Child 2004, 89:125-30.

Dated: 29th Sept, 2016

- 13. Cortesi F, Giannotti F, Ivanenko A, Johnson K: Sleep in children with autistic spectrum disorder. Sleep Med 2010, 11:659-64.
- 14. Weiss MD, Wasdell MB, Bomben MM, Rea KJ, Freeman RD. Sleep hygiene and melatonin treatment for children and adolescents with ADHD and initial insomnia. Journal of the American Academy of Child & Adolescent Psychiatry. 2006; 45(5):512-9.
- Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep 2000; 23(8):1043-1051.
- 16. Tso K. Sleep. Masters thesis. Department of Community Medicine: The Chinese University of Hong Kong. 2001.
- 17. Drake, C., Nickel, C., Burduvali, E., Roth, T., Jefferson, C., & Badia, P. (2003). The pediatric daytime sleepiness scale (PDSS): sleep habits and school outcomes in middle-school children. SLEEP-NEW YORK THEN WESTCHESTER-, *26*(4), 455-460.
- 18. Yang, C. M., Huang, Y. S., & Song, Y. C. (2010). Clinical utility of the Chinese version of the Pediatric Daytime Sleepiness Scale in children with obstructive sleep apnea syndrome and narcolepsy. Psychiatry and clinical neurosciences, 64(2), 134-140.
- 19. Meltzer LJ, Westin AM. A comparison of actigraphy scoring rules used in pediatric research. Sleep Med 2011;12:793-6.
- 20. American Psychiatric Association (1994), Diagnosite and Statistical Manual of Mental Disorders, 4th edition (DSM-IV). Washington, DC: American Psychiatric Association.
- 21. Ho TP, Leung PWL, Lee CC, Tang CP, Hung SF, Kwong SL, Lucas CP, Lieh-Mak F, Shaffer D. (2005) Test-retest reliability of the Chinese version of the Diagnostic Interview Schedule for Children-Version 4 (DISC-IV). J of Child Psycho and Psychiat. 46,10, 1135-1138.
- 22. Shaffer D. Fisher P, Lucas C, Dulcan M, Schwab-Stone M. NIMH Diagnostic Interview Schedule for Children Version IV (NIMH DISC-IV): description, differences from previous versions, and reliability of some common diagnoses. J Am Acad Child Adolesc Psychiatry 2000; 39:28-38.
- 23. Lai KY, Leung PW, Luk ES, Wong AS, Law LS, Ho KK. Validation of the Chinese strengths and weaknesses of ADHD-symptoms and normal-behaviors questionnaire in Hong Kong. Journal of attention disorders. 2013;17(3):194-202.
- 24. Achenbach, T. M., & Rescorla, L. (2001). ASEBA school age forms & profiles.
- 25. Leung PW, Kwong SL, Tang CP et al. Test-retest reliability and criterion validity of the Chinese version of CBCL, TRF, and YSR. J Child Psychol Psychiatry 2006; 47(9):970-973.
- 26. Varni J, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr 2003; 3:329-41.

Dated: 29th Sept, 2016

- 27. Goodman, R. Psychometric properties of the Strengths and Difficulties Questionnaire (SDQ). J Am Acad Child Adolesc Psychiatry. 2001; 40(11): 1337-1345.
- 28. Lai, K. Y., Luk, E. S., Leung, P. W., Wong, A. S., Law, L., and Ho, K. Validation of the Chinese version of the strengths and difficulties questionnaire in Hong Kong. Soc Psychiatry Psychiatr Epidemiol. 2010; 45(12): 1179-86.
- 29. Mueller, S. T., & Piper, B. J. (2014). The Psychology Experiment Building Language (PEBL) and PEBL Test Battery. Journal of Neuroscience methods.
- 30. Mueller, S. T. (2011). The PEBL digit span test. Computer software retrieved from http://pebl.sf.net/battery.html
- 31. Mueller, S. T. (2011). The PEBL n-back test. Computer software retrieved from http://pebl.sf.net/battery.html
- 32. Mueller, S. T. (2011). The PEBL Digit letter test. Computer software retrieved from http://pebl.sf.net/battery.html
- 33. Mueller, S. T. (2011). PEBL's Berg Card Sorting Test-64 (PBCST-64) Computer software retrieved from http://pebl.sf.net/battery.html
- 34. Mueller, S. T. (2011). The PEBL Tower of London Test. Computer software retrieved from http://pebl.sf.net/battery.html
- 35. Shallice, T. (1982). Specific impairments of planning. Philosophical Transactions of the Royal Society of London. Series B, Biological Sciences. 298(1089): 199–209.
- 36. Buysse, D. J., Reynolds, C. F., Monk, T. H., Berman, S. R., & Kupfer, D. J. (1989). The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry research, 28(2), 193-213.
- 37. Tsai PS, Wang SY, Wang MY, et al. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res 2005; 14:1943-52.
- 38. Bastien CH, Vallières A, Morin CM. Validation of the insomnia severity index as an outcome measure for insomnia research. Sleep medicine 2 2001; 297-307.
- 39. Chung, K. F., Kan, K. K., & Yeung, W. F. (2011). Assessing insomnia in adolescents: Comparison of insomnia severity index, Athens insomnia scale and sleep quality index. Sleep Medicine, 12(5), 463-470.
- 40. Mastin, D.F., Bryson, J. & Corwyn, R. J Behav Med (2006) 29: 223. doi:10.1007/s10865-006-9047-6
- 41. Johns, M. W. (1994). Sleepiness in different situations measured by the Epworth Sleepiness Scale. SLEEP-NEW YORK-, 17, 703-703.

Dated: 29th Sept, 2016

- 42. Chung, KF. (2000). Use of the Epworth Sleepiness Scale in Chinese patients with obstructive sleep apnea and normal hospital employees. J Psychosom Res. 49(5):367–372.
- 43. Abidin, R. R. (1990). Parenting stress index-short form. Charlottesville, VA: Pediatric Psychology Press.
- 44. Tam KK, Chan YC, Wong CKM. Validation of the parenting stress index among Chinese mothers in Hong Kong. Journal of Community Psychology 1994; 22(3):211-223.
- 45. Lovibond PH, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther 1995; 33:335-43.
- 46. Taouk M, Lovibond P, Laube R. Psychometric properties of a Chinese version of the 21-item Depression Anxiety Stress Scales (DASS21). Report for New South Wales Transcultural Mental Health Centre, Cumberland Hospital, Sydney. 2001.
- 47. Smets, E. M. A., Garssen, B., Bonke, B. D., & De Haes, J. C. J. M. (1995). The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. Journal of psychosomatic research, 39(3), 315-325.
- 48. Chung, K. F., Yu, B. Y. M., Yung, K. P., Yeung, W. F., Ng, T. H., & Ho, F. Y. Y. (2014). Assessment of fatigue using the Multidimensional Fatigue Inventory in patients with major depressive disorder. Comprehensive psychiatry, 55(7), 1671-1678.
- 49. Hiscock, H., Sciberras, E., Mensah, F., Gerner, B., Efron, D., Khano, S., & Oberklaid, F. (2015). Impact of a behavioural sleep intervention on symptoms and sleep in children with attention deficit hyperactivity disorder, and parental mental health: randomised controlled trial. BMJ, 350, h68.
- 50. Barnett AG, van der Pols JC, Dobson AJ. Regression to the mean: what it is and how to deal with it. Int J Epidemiol. 2005;34(1):215–220).
- 51. Cohen, J. (1992). A power primer. Psychological bulletin, 112(1), 155.

Dated: 29th Sept, 2016

# Appendix

Figure 1.



Dated: 29<sup>th</sup> Sept, 2016 Version number: 1.2 – Clincial Trial Registration

## Recruitment criteria (for psychiatrists' reference):

### Inclusion criteria:

- 6-12 years old (of both genders)
- ADHD (any subtype)
- With insomnia (difficulty initiating and/or maintaining sleep)

## Excluding those with the following condition

- Serious medical condition (e.g. severe cerebral palsy) or intellectual disability (IQ<70)
- Neurological and/or medical condition that may lead to disordered sleep
- Clinical sleep disorders (e.g. obstructive sleep apnea, OSA)
- Receiving specialized help (behavioural intervention) for their sleep from a psychologist or at a specialized sleep clinic

Dated: 29th Sept, 2016